CLINICAL TRIAL: NCT02595580
Title: An Open, Controlled Investigation of Measurement Precision, System Accuracy and User Performance Evaluation in Subjects With Diabetes Mellitus Type 1 Using GlucoPred, a Non-invasive Continuous Blood Glucose Measurement Device
Brief Title: The GlucoPred Investigation II
Acronym: GPI-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: skin irritation caused by device
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset Ostfold (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-GPI-II-2015
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Blood Glucose Self-Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GlucoPred (Experimental)
  Interventions: Device: Glucopred

INTERVENTIONS:
Device: Glucopred

SUMMARY:
Diabetes mellitus type 1 (DM1) is an autoimmune metabolic disease in which the insulin producing cells in the pancreas are destroyed and the subject is left totally dependent of external supply of insulin. There is no known cure for DM1 except for in very specific situations. Thus, management of DM1 concentrates on keeping blood glucose levels as close to normal levels.

As an aid to subjects with DM1 for managing their blood glucose levels as close to normal as possible, blood glucose monitoring systems have been developed. Available blood glucose monitoring systems today require a capillary blood sample that is analysed by a glucose meter. Subjects are normally advised by health care professionals on the appropriate blood glucose monitoring regime for their condition. However, many subjects fail to measure blood glucose as often as needed to achieve good blood glucose control despite every effort from health care professionals.

Research and development of non-invasive interstitial blood glucose monitoring methods is ongoing. All attempts to develop a non-invasive continuous glucose measuring device have so far failed. Prediktor Medical AS has developed a non-invasive sensor, GlucoPred, based on the combination of several non-invasive measurement principles and multivariate analysis and dynamic models of glucose/insulin interaction. The device will be body mounted in the form of a bracelet or a watch communicating with a mobile phone or a tablet for data presentation and collection. Development of GlucoPred is now at a stage where testing of the sensor in subjects under controlled settings is required before further development can take place.

If successful, this will be a major step ahead for all patients with diabetes and markedly increase their possibility to take care of their disease on a day to day basis without the burden of frequent blood sampling or wearing an invasive device.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 1
* has read and understood the informed consent documentation and is willing to participate in the investigation and willing to sign the informed consent form
* willing to participate in the investigation using one or two GlucoPred sensors for a period of 8 days
* willing to attend 2 investigational visits with duration of up to 4 hours during the investigational period
* willing to take and record up to 16 finger-stick blood samples on Day 1 and up to 8 finger-stick blood samples daily for measuring reference values for the duration of the investigation
* Uses a blood-glucose monitoring system for self-testing on a daily basis
* Willing to use the provided blood-glucose monitoring system during the investigation
* Has access to and is willing to use a computer for downloading data and charging the sensor

Exclusion Criteria:

* not fit for the investigation due concurrent illness
* Unfit for participation for any reason judged by the investigator
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
difference between Glucopred and the reference method | 8 days
  degree of point and trend accuracy between GlucoPred measured values and values measured by the reference methods

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, md prof, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Sykehuset Østvold, Fredrikstad
  - St Olavs Hospital, Trondheim